CLINICAL TRIAL: NCT02536430
Title: Efficacy of Ketorolac Buccal Infiltration on Success Rate of Inferior Alveolar Nerve Block in Patients With Irreversible Pulpitis: A Prospective, Randomized, Double-blind Clinical Trial
Brief Title: Efficacy of Ketorolac Buccal Infiltration on Success Rate of Inferior Alveolar Nerve Block
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nahid Mohammadzadeh Akhlaghi (Other)
Responsible Party: Sponsor-Investigator, Nahid Mohammadzadeh Akhlaghi, Doctor Nahid Mohammadzadeh Akhlaghi, Azad University of Medical Sciences
Organization: Azad University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AZadUMS-P/212/D
Record Dates: First submitted 2015-08-21; First posted 2015-08-31 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Failed Mechanical Induction
Keywords: Infra alveolar nerve block; Ketorolac; Success rate
MeSH Terms: interventions — Ketorolac Tromethamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buccal infiltration of Ketorolac (Active Comparator): A buccal infiltration of 30 mg/mL of Ketorolac Tromethamine was applied for the patients in case group.
  Interventions: Drug: Ketorolac Tromethamine
- buccal infiltration of Normal Saline (Placebo Comparator): A buccal infiltration of Normal Saline was applied for the patients in control group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac Tromethamine — One group received a buccal infiltration of Ketorolac Tromethamine
  Other Names: Toradol
  Arms: Buccal infiltration of Ketorolac
Drug: Placebo — buccal infiltration of Normal Saline.
  Other Names: Normal Saline
  Arms: buccal infiltration of Normal Saline

SUMMARY:
The aim of this study was to determine whether combining an intraoral injection of a non steroidal anti-inflammatory drug (Ketorolac), in association with conventional inferior alveolar nerve block, would improve the success rate in teeth with irreversible pulpitis. Forty adult volunteers with including criteria has been randomly divided into two groups (n=20). All patients received standard inferior alveolar nerve block injection. After achieving the lip numbness, one group received a buccal infiltration of Ketorolac and the other one received a buccal infiltration of Normal Saline as placebo. Any pain during root canal treatment has been recorded using analog visual scale. The success was considered as none or mild pain during treatment. The data have been analyzed using Mann-U-Whitney and chi-squared tests.

DETAILED DESCRIPTION:
Objectives:

The aim of this study was to determine whether combining an intraoral injection of a non steroidal anti-inflammatory drug (Ketorolac), in association with conventional inferior alveolar nerve block, would improve the success rate in teeth with irreversible pulpitis.

Design: Randomized double blind clinical trial

Setting and conduct: Forty adult volunteers will randomly divide into two groups (n=20). All patients will receive standard inferior alveolar nerve block injection of 4% Articaine with 1:100000 epinephrine and supplemental buccal infiltration of 0.9 mL 4% Articaine with 1:100000 epinephrine. After five minutes when the lip numbness was achieved, one group received supplemental buccal infiltration of 30 mg/mL of Ketorolac Tromethamine and other group received buccal infiltration of normal saline. Endodontic access preparation initiated after 15 minutes of initial IANB with two negative responses to the electric pulp test. Pain during caries and dentin removal, access cavity preparation and canal length measurements has been recorded using visual analog scale (VAS). The success was considered as none or mild pain during the treatment. The data have been analyzed using Mann-U-Whitney and chi-squared tests.

Participants including major eligibility criteria: all patients with symptomatic irreversible pulpitis (Heft Parker VAS ≥54) of a mandibular molar tooth without systemic diseases; non smoking; without any medicine consumption or analgesic and sedation Intervention: Ketorolac infiltration

Main outcome measures : Pain during caries and dentin removal , access cavity preparation and canals length measurements using VAS.

ELIGIBILITY:
Inclusion Criteria:

* patients with age ranged 18-65;
* without systemic diseases;
* without any medicine consumption;
* non smoking;
* non pregnant;
* non breast feeding;
* with symptomatic irreversible pulpitis (Visual Analog Scale ≥ 54) in one mandibular molar that needs root canal treatment

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of Ketorolac infiltration on success rate of inferior alveolar nerve block | One week

CONTACTS AND LOCATIONS:
Overall Officials: Nahid Mohammadzadeh Akhlaghi, DDS,MDS, Principal Investigator — Associate Professor
Locations (1):
- Dental Branch, AZad UMS, Tehran, Tehran Province, Iran